CLINICAL TRIAL: NCT00645697
Title: Intravitreal Bevacizumab in Recalcitrant Inflammatory Ocular Neovascularization: Multicenter Collaborative Study
Brief Title: Intravitreal Bevacizumab in Recalcitrant Inflammatory Ocular Neovascularization
Acronym: AVA-ION
Status: Completed | Type: Observational
Sponsor: Rafic Hariri University Hospital (Other)
Collaborators: Heidelberg University (Other); University Hospital Tuebingen (Other); University Hospital Freiburg (Other)
Responsible Party: Ahmad Mansour, AUB
Other Study IDs: 1955AM
Record Dates: First submitted 2008-03-25; First posted 2008-03-28 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Neovascularization; Tuberculosis; Multifocal Serpiginous Choroiditis; Harada Toxoplasmosis
Keywords: tuberculosis; Multifocal serpiginous choroiditis; histoplasmosis; Harada toxoplasmosis
MeSH Terms: conditions — Neovascularization, Pathologic; Tuberculosis; Histoplasmosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
One complication of uveitis which is driven by an increase in VEGF is the formation of inflammatory ocular neovascularization (ION). Here, we analyze the therapeutic role of intravitreal bevacizumab in ION not responding to standard therapy (systemic and ocular corticosteroids and systemic immunosuppressants) in a multicenter retrospective study.The natural history of subfoveal choroidal new vessels histoplasmosis, multifocal choroiditis, Harada and other inflammatory chorioretinal disorders has been very guarded, but with this new approach, we hope to stop the visual loss in these relatively young patients.

DETAILED DESCRIPTION:
Members of the American Society of Retinal specialists, the American Uveitis Society and the International Uveitis Society were invited to contribute their consecutive cases of ION not responding to standard therapy (corticosteroids (CST) 4 or immunosuppression) and treated with intravitreal anti-VEGF agents. Cases with concomitant or prior cystoid macular edema, diabetes mellitus, or age-related macular degeneration were excluded. Most of the patients had initially been treated in a stepwise fashion with high doses of oral CST, with or without intraocular or subtenon CST or immunosuppressive therapy (as monitored by a rheumatologist). All patients opted to intravitreal anti-VEGF treatment after detailed information about the limited experience, potential side effects and the off-label character of the drug. The risks and benefits of intravitreal therapy were discussed with the patients (or their guardians) who signed an informed consent. Primary outcome measure: Best corrected visual acuity measured as logMAR. Secondary outcome measures:macular thickness on OCT, and stoppage of leakage by IVFA.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory ocular neovascularization (INO)

Exclusion Criteria:

* Eyes with age-related macular degeneration
* Diabetes mellitus
* Prior cystoid macular edema
* Uncontrolled systemic hypertension
* Cardiovascular disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective review of INO treated by the 25 collaborators from the 5 continents.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2007-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Best corrected visual acuity gain after bevacizumab therapy. | 3 month, 1 year, 2 year

SECONDARY OUTCOMES:
fluorescein leakage of ocular neovascularization by fluorescein angiography and macular thickness by Optical Computed tomography. | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M Mansour, MD, Principal Investigator — American University of Beirut Rafic Hariri University Hospital
Locations (1):
- American University of Beirut, Beirut, Lebanon

REFERENCES:
- [Derived] Mansour AM, Arevalo JF, Fardeau C, Hrisomalos EN, Chan WM, Lai TY, Ziemssen F, Ness T, Sibai AM, Mackensen F, Wolf A, Hrisomalos N, Heiligenhaus A, Spital G, Jo Y, Gomi F, Ikuno Y, Akesbi J, LeHoang P, Adan A, Mahendradas P, Khairallah M, Guthoff R, Ghandour B, Kucukerdonmez C, Kurup SK. Three-year visual and anatomic results of administrating intravitreal bevacizumab in inflammatory ocular neovascularization. Can J Ophthalmol. 2012 Jun;47(3):269-74. doi: 10.1016/j.jcjo.2012.03.042. PMID 22687305
- [Derived] Mansour AM, Arevalo JF, Ziemssen F, Mehio-Sibai A, Mackensen F, Adan A, Chan WM, Ness T, Banker AS, Dodwell D, Chau Tran TH, Fardeau C, Lehoang P, Mahendradas P, Berrocal M, Tabbarah Z, Hrisomalos N, Hrisomalos F, Al-Salem K, Guthoff R. Long-term visual outcomes of intravitreal bevacizumab in inflammatory ocular neovascularization. Am J Ophthalmol. 2009 Aug;148(2):310-316.e2. doi: 10.1016/j.ajo.2009.03.023. Epub 2009 May 9. PMID 19427992
- [Derived] Mansour AM, Mackensen F, Arevalo JF, Ziemssen F, Mahendradas P, Mehio-Sibai A, Hrisomalos N, Lai TY, Dodwell D, Chan WM, Ness T, Banker AS, Pai SA, Berrocal MH, Tohme R, Heiligenhaus A, Bashshur ZF, Khairallah M, Salem KM, Hrisomalos FN, Wood MH, Heriot W, Adan A, Kumar A, Lim L, Hall A, Becker M. Intravitreal bevacizumab in inflammatory ocular neovascularization. Am J Ophthalmol. 2008 Sep;146(3):410-416. doi: 10.1016/j.ajo.2008.05.024. Epub 2008 Jul 10. PMID 18619571